CLINICAL TRIAL: NCT00720421
Title: A Phase 1, Single Centre, Single Dose, Double-blind, Double-dummy, Four-way Crossover, Placebo-controlled, Randomized Study to Investigate the Effects of AZD7325 on Sedation, Cognition and Electroencephalogram (EEG) in Comparison With Lorazepam in Healthy Male Volunteers.
Brief Title: A Sedation/Cognition/Electroencephalogram (EEG) Study Using AZD7325 and Comparator.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Smith, MD, Medical Science Director, Emerging Psychiatry, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1140C00003; EudractCT 2008-001757-17
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-11

CONDITIONS: Healthy Volunteer
Keywords: Phase I; pharmacodynamic study
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Other): AZD7325 Placebo/Lorazepam Placebo combination therapy; washout period; AZD7325 10 mg/Lorazepam Placebo combination therapy; washout period; AZD7325 Placebo/Lorazepam 1 mg combination therapy; washout period; AZD7325 1 mg/Lorazepam Placebo combination therapy
  Interventions: Drug: AZD7325; Drug: Lorazepam
- 2 (Other): AZD7325 10 mg/Lorazepam Placebo combination therapy; washout period; AZD7325 1mg/Lorazepam Placebo combination therapy; washout period; AZD7325 Placebo/Lorazepam Placebo combination therapy; washout period; AZD7325 Placebo/Lorazepam 1 mg combination therapy
  Interventions: Drug: AZD7325; Drug: Lorazepam
- 3 (Other): AZD7325 Placebo/Lorazepam 1 mg combination therapy; washout period; AZD7325 Placebo/Lorazepam Placebo combination therapy; washout period; AZD7325 1 mg/Lorazepam Placebo combination therapy; washout period; AZD7325 10 mg/Lorazepam Placebo combination therapy
  Interventions: Drug: AZD7325; Drug: Lorazepam
- 4 (Other): AZD7325 1 mg/Lorazepam Placebo combination therapy; washout period; AZD7325 Placebo/Lorazepam 1 mg combination therapy; washout period; AZD7325 10 mg/Lorazepam Placebo combination therapy; washout period; AZD7325 Placebo/Lorazepam Placebo combination therapy
  Interventions: Drug: AZD7325; Drug: Lorazepam

INTERVENTIONS:
Drug: AZD7325 — AZD7325 10 mg oral 2 capsules
Drug: AZD7325 — AZD7325 1 mg oral 2 capsules
Drug: AZD7325 — AZD7325 Placebo oral 2 capsules
Drug: Lorazepam — Lorazepam 1 mg oral 2 tablets
Drug: Lorazepam — Lorazepam Placebo oral 2 tablets

SUMMARY:
The purpose of the study is to determine the effects of the compound AZD7325 as compared to lorazepam on sleepiness, concentration and brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged 18 to 55 years on screening

Exclusion Criteria:

* Clinically significant illness within 2 weeks before the study start
* Enrollment in another concurrent investigational study or intake of an investigational drug within 30 days or intake of an investigational drug within a period of 5 half lives of that drug prior to the screening visit
* Blood loss in excess of 200 mL within 30 days of Day -2, in excess of 400 mL within 90 days of Day -2, or in excess of 1200 mL within 1 year of Day -2
* Clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacodynamic effects of AZD6280 by central nervous system function tests. | Test batteries will be performed at specified times both before and following study drug administration.

SECONDARY OUTCOMES:
Evaluation and characterization of the pharmacokinetics of AZD6280. | Blood samples will be taken during the study.

CONTACTS AND LOCATIONS:
Overall Officials: J.M.A. Van Gerven, MD, PhD, Principal Investigator — CHDR Leiden, the Netherlands
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands